CLINICAL TRIAL: NCT04041336
Title: Optical Coherence Tomography Feasibility in Older People Following Hip Fracture Surgery
Brief Title: Hand-held Optical Coherence Tomography Feasibility Older Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19006
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Retinal Imaging
Keywords: Older; Hip fracture surgery; Optical coherence tomography
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Assess the feasibility of measuring the thickness of retinal layers using a handheld optical coherence tomography device in older patients after hips fracture surgery. Consecutively recruited consenting patients will be included.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will have measurements taken. There are no comparators or controls in this feasibility study
  Interventions: Diagnostic Test: Optical coherence tomography

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography — Non-invasive method of acquiring cross sectional imaging of tissues using the coherent property of light
  Other Names: OCT

SUMMARY:
Assessment of the feasibility of achieving retinal imaging in older people with recent hips fracture surgery using hand held optical coherence tomography device

DETAILED DESCRIPTION:
Optical coherent tomography (OCT) is a device used to achieve cross-sectional imaging of tissues. It is often used in ophthalmology and also has application in dermatology, cardiology and other specialities. Usually, in adults, a table-top device is used necessitating the transfer of patients to the location of the device. In children a hand held device is used meaning the device can be taken to the patients' location. To facilitate/ help design a future study, this study's aim is to assess the feasibility of achieving retinal imaging in older people who are recovering from hip fracture surgery using a hand held device.

ELIGIBILITY:
Inclusion Criteria:

* Recent hip fracture surgery
* Age > 64 years
* No cognitive impairment
* Able to understand instructions given in English
* Consent

Exclusion Criteria:

* Presence of degenerative eye disease e.g. age-related macula degeneration, glaucoma, diabetic retinopathy, hypertensive retinopathy
* Dementia, mild cognitive impairment, Parkinson,s disease, multiple sclerosis, current delirium

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Ability to achieve good quality retinal images | 30 minutes
  Retinal images with signal strength > 6 and in which retinal layers can be measured
Ability to achieve imaging without causing pain | Immediate
  Patient reported pain during acquisition of images over their baseline. Scale of 0 - 10 where 0 is no increase in pain and 10 is severe increase in pain

CONTACTS AND LOCATIONS:
Overall Officials: Iain Moppett, PhD, Principal Investigator — University of Nottingham, Nottingham, UK
Locations (1):
- Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data on our primary outcome will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date 6 months after publication. End date 12 months after publication
Access Criteria: Researchers with a valid reason as reviewed by the lead investigator